CLINICAL TRIAL: NCT04152473
Title: Phase 1 Study to Test Safety and Dose of Proglumide as an Anti-fibrotic Agent in Non-alcoholic Steatohepatitis (NASH)
Brief Title: Safety and Tolerability of Oral Proglumide for NASH
Acronym: STOPNASH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 0562; GU-3160 (Other: Georgetown University)
Record Dates: First submitted 2019-10-20; First posted 2019-11-05 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Nonalcoholic Steatohepatitis
Keywords: NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Proglumide

STUDY DESIGN:
Intervention Model Description: open labelled sequential Phase I ascending dose study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Proglumide (Experimental): Open labelled proglumide treated
  Interventions: Drug: Proglumide

INTERVENTIONS:
Drug: Proglumide — oral CCK receptor antagonist
  Other Names: Milid

SUMMARY:
This study is an open labelled Phase I/II clinical trial, designed to evaluate the safety and efficacy of an oral cholecystokinin (CCK) receptor antagonist, proglumide, at escalating doses in subjects with NASH.

An extended use protocol has been approved for subjects completing this study that show benefit or are at risk of Liver disease progression to continue on Proglumide at 1200 mg / day for an additional 3-9 months. Subjects in the extended protocol will have telephone visits monthly and in the research unit every 3 months for safety lab tests and research blood for fibrosis analysis.

DETAILED DESCRIPTION:
This is a Phase 1single ascending dose study in 18 patients with ultrasound evidence of fatty liver disease AND increased hepatic transaminases. Proglumide will be using the single ascending dose study design in a Phase 1 fashion to determine the recommended Phase 2 dose (RP2D). Dose levels of proglumide will be: 400mg BID (twice daily); 400 mg TID (three times daily); 800 mg BID (twice daily).

Six patients will be enrolled in each cohort starting with the lowest dose of 400mg po BID (Twice daily)for 12 weeks.

Patients will be monitored for safety and toxicity by laboratory blood testing, physical examinations. Blood level for proglumide will be done at before proglumide at screening or baseline, week 2 and then week 4 and week 12.

Safety and toxicity will be monitored using the Common Terminology Criteria for Adverse Events v 5 and 'efficacy 'of the treatment will be evaluated by assessment of liver enzymes and fibroscan. The Phase 1 study design, we will follow the dose escalation scheme, where the dose increases after 6 subjects if a drug limiting toxicity (DLT) does not occur.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ages 18 years to 85
* with radiographic imaging (by ultrasound, MRI, or CT) of fatty liver disease
* AND elevation in serum transaminases (ALT or AST).
* AND one of the following: BMI>30, hyperlipidemia, or evidence of poorly controlled diabetes such as HgbA1C >7
* Subjects on statins and with diabetes are eligible. Statins will be continued at the same dose for the duration of the study.
* Evidence of mild to moderate fibrosis on Fibroscan of F1 to F3 (kPa score < 14).

Exclusion Criteria:

* Evidence of active alcohol use/abuse.
* Chronic viral hepatitis B or hepatitis C, autoimmune hepatitis, drug induced liver disease.
* Those with evidence of cirrhosis on exam, histologically, or imaging, and a history of liver cancer are excluded.
* Laboratory tests that warrant exclusion include: Leukocyte Count <3.5 K/UL; Hemoglobin <9.5 g/dL; Blood Urea Nitrogen >30 mg/dL (hydrated); Creatinine >2.0 mg/dL, alanine aminotransferase (ALT)/ aspartate aminotransferase (AST) > 5X ULN (upper limit normal), alkaline phosphatase (ALP)>2X ULN.
* Evidence of abnormal synthetic liver function including abnormal total bilirubin, platelet count <150,000 / mm3; and abnormal prothrombin time or increased INR (international normalized ratio) (unless on warfarin)
* History of gall bladder disease with gall bladder not surgically removed
* Estimated glomerular filtration rate (eGFR of < 90 mL/min/1.73m2
* Type 1 diabetes mellitus
* Poorly controlled diabetes, defined by hemoglobin A1C (HbA1C) > 8, or diabetic patients that have not been on stable doses of anti-diabetic medication for at least 90 days prior to screening
* Pregnant or breast feeding
* A known preexisting medical or psychiatric condition that could interfere with the patient's ability to provide informed consent or participate in study conduct, or that may confound the study findings.

  * Those found to have fibrosis score on Fibroscan of F0 or F4.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
safety and toxicity | 12-weeks per dose
  Number of participants with drug related Toxicity will follow standard Common Terminology Criteria for Adverse Events v.5,(CTCAE) criteria protocols. Toxicity is graded according to severity for symptoms obtained on the visit review of symptoms and according to blood tests collected at each scheduled visit
Recommended Phase 2 dose | for each dose, the number of AEs described over the 12 week period
  Of the 3 doses to be tested which one has the fewest Drug related toxicity

SECONDARY OUTCOMES:
Liver transaminases | Comparison of baseline serum ALT and AST values to week 12 week values in IU
  A decrease in the serum aminotransferases (ALT and AST) in IU by 10% or more

OTHER OUTCOMES:
NASH score by Fibroscan | baseline compared to week 12
  liver stiffness kPa score with a decrease by 4kPa and steatosis (CAPS) score in dB/m. a decline of 30 dB/m

CONTACTS AND LOCATIONS:
Overall Officials: Jill P Smith, MD, Principal Investigator — Georgetown University
Locations (2):
- United States (2):
  - Georgetown University, Washington D.C., District of Columbia
  - Washington DC Veterans Affairs Medical Center, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: Yes
The data will be uploaded on the clinical trials website at the conclusion of the study and after accepted for publication
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After the publication at the completion of the study
Access Criteria: Available on clinicaltrials.gov website for 1 year after publication

REFERENCES:
- [Background] Tucker RD, Ciofoaia V, Nadella S, Gay MD, Cao H, Huber M, Safronenka A, Shivapurkar N, Kallakury B, Kruger AJ, Kroemer AHK, Smith JP. A Cholecystokinin Receptor Antagonist Halts Nonalcoholic Steatohepatitis and Prevents Hepatocellular Carcinoma. Dig Dis Sci. 2020 Jan;65(1):189-203. doi: 10.1007/s10620-019-05722-3. Epub 2019 Jul 11. PMID 31297627
- [Background] Rabiee A, Gay MD, Shivapurkar N, Cao H, Nadella S, Smith CI, Lewis JH, Bansal S, Cheema A, Kwagyan J, Smith JP. Safety and Dosing Study of a Cholecystokinin Receptor Antagonist in Non-alcoholic Steatohepatitis. Clin Pharmacol Ther. 2022 Dec;112(6):1271-1279. doi: 10.1002/cpt.2745. Epub 2022 Sep 27. PMID 36087237